CLINICAL TRIAL: NCT05393141
Title: The Effect of Body Weight Management and Cognitive Exercise Therapy Approach on Psoriatic Arthritis Symptoms
Brief Title: The Effects of Weight Loss on Psoriatic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sumeyra Oteles, Clinical Researcher of the Hacettepe University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HU-SO-2022
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Psoriatic Arthritis; Obesity
Keywords: psoriatic arthritis; diet; biopsychosocial exercise
MeSH Terms: conditions — Arthritis, Psoriatic; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- diet group (Experimental): weight loss diet intervention for 12 weeks
  Interventions: Behavioral: diet and biopsychosocial exercise intervention
- diet+bety group (Experimental): weight loss diet intervention for 12 weeks and exercise-based biopsychosocial approach (Cognitive Exercise Therapy Approach-BETY) intervention for 12 weeks
  Interventions: Behavioral: diet and biopsychosocial exercise intervention
- control group (No Intervention): no intervention, control

INTERVENTIONS:
Behavioral: diet and biopsychosocial exercise intervention — dietary intervention: biopsychosocial exercise intervention:
  Arms: diet group; diet+bety group

SUMMARY:
Psoriatic arthritis (PsA) is an inflammatory arthritis associated with psoriasis. Although the underlying cause of PSA is unclear, increased body weight is known to increase the disease symptoms. This study aims to determine the effects of dietary and Cognitive Exercise Therapy Approach (BETY-Bilişsel Egzersiz Terapi Yöntemi) interventions on symptoms. Accordingly, 45 overweight/obese subjects with PSA aged 20-65 years will divide into "diet", "diet+bety", and "control" groups. Dietary, laboratory and anthropometric records, Short Form Health Survey, DAPSA (Disease Activity in Psoriatic Arthritis), HAQ (Health Assesment Questionnaire) of all subjects will compare at the baseline and at the end of the study.

DETAILED DESCRIPTION:
Although the underlying cause of PSA is unclear, increased body weight is known to increase the disease symptoms. The present study aims to determine the effects of dietary and Cognitive Exercise Therapy Approach interventions on symptoms.

* Fourt-five overweight/obese subjects with PSA aged 20-65 years will divide into diet (n=15), diet+bety (n=15), and control (n=15) groups.
* Individually diet programs will be applied according to the metabolic, biochemical, and physical activity status of the subjects prepared by a registered dietitian.
* BETY exercise training will be given by a registered physiotherapist.
* The subjects will be followed for 12 weeks.
* Dietary, laboratory and anthropometric records, Short Form Health Survey, DAPSA (Disease Activity in Psoriatic Arthritis), HAQ (Health Assesment Questionnaire) of all subjects will compare at the baseline and at study completion.

ELIGIBILITY:
Inclusion Criteria:

* overweight/obese
* diagnosed with PSA

Exclusion Criteria

* pregnancy or lactation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Weight Loss | At the end of 3 months
  BMI (kilogram/metre2(kg/m2))
DAPSA score | At the end of 3 months
  The score ranges from 0 to 50 points, with increased score reflect more discomfort

SECONDARY OUTCOMES:
Quality of Life Score | At the end of 3 months
  The score ranges from 0 to 100 points, with increased score reflecting improved quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Sümeyra Öteleş, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No